CLINICAL TRIAL: NCT00005571
Title: A Randomized, Third-Party-Blind, Placebo-Controlled Pilot Study of the Effect of h5G1.1-mAb on Dermatomyositis Patients
Brief Title: Safety and Effectiveness of h5G1.1-mAb for Dermatomyositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000117; 00-AR-0117
Record Dates: First submitted 2000-04-25; First posted 2000-04-26 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-12

CONDITIONS: Dermatomyositis
Keywords: Skin; Humoral Immunity; Myositis; Complement; Antibody; Dermatomyositis
MeSH Terms: conditions — Dermatomyositis; Myositis

INTERVENTIONS:
Drug: h5G1.1-mAb

SUMMARY:
This study will evaluate the safety and effectiveness of the experimental drug h5G1.1-mAb in treating patients with dermatomyositis. This disease, which causes skin rash, muscle weakness, and sometimes various other symptoms, may be due to an immune system abnormality. Drugs currently used to treat dermatomyositis, such as prednisone and various anticancer drugs, often have serious side effects and may not work in all patients. h5G1.1-mAb is a genetically engineered antibody that blocks the activity of certain proteins involved in the immune reaction that produces inflammation.

Patients age 18 years and older who have had dermatomyositis for at least 6 months and who have not improved with prednisone or other therapies, or who cannot tolerate prednisone or other therapies, may be eligible for this 12-week study. Candidates will have a history and physical examination, including blood and urine tests, throat culture, and muscle strength testing. Participants will be randomly assigned to receive either h5G1.1-mAb or placebo (an inactive substance). The drug or placebo will be given intravenously (through a thin tube inserted into a vein) once a week for five doses and then every other week for two more doses.

Participants will undergo the following additional tests at various intervals during the study as follows:

1. Complete physical examination ( visit 9)
2. Blood and urine tests (various intervals)
3. Muscle strength testing, assessment of ability to perform daily tasks, and completion of questionnaire regarding functional abilities (visits 2, 6 and 9)
4. Ultrasound imaging of muscle (during certain muscle exercises) (visits 2, 6 and 9)
5. Electrocardiogram (EKG) (visits 2 and 9)
6. Throat swab (culture) (visit 6)
7. Examination and photography of skin lesions (visits 2 and 9)
8. Skin biopsy - removal of small sample of skin tissue under local anesthetic (visits 2 and 9)
9. Magnetic resonance imaging (MRI) scan of muscles (visits 2 and 9)
10. Possible muscle biopsy - removal of small sample of muscle tissue under local anesthetic (visits 2 and 9).

DETAILED DESCRIPTION:
This is a randomized, third-party, placebo-controlled pilot study of h5G1.1-mAb, an antibody directed at the complement component C5, administered to patients with dermatomyositis with persistent disease. We are one of the four groups taking part in a multicenter trial under the sponsorship of Alexion Pharmaceuticals, Inc.

In dermatomytosis, humorally-mediated damage to muscle and skin microvasculature appears very important. The deposition of the membrane attack complex (C5-9) on the capillaries has been shown to precede the destruction of muscle fibers and to be a specific finding in the skin lesion. These observations, along with the recent discovery of the effectiveness of intravenous gammaglobulin (IVIG) in dermatomyositis, support the role of complement activation in the pathogenesis of dermatomyositis. Among the activated components of the complement system, the products that are generated after cleavage of C5, namely, C5a and C5b-9, are potent inflammatory mediators with pleiotropic activities. Inhibition of complement activation at C5 would prevent the formation of these pro-inflammatory molecules while allowing the generation of C3b, which is critical for opsonization and immune complex clearance. C5 inhibition therefore represents a potentially effective therapeutic modality for dermatomyositis.

Anti-C5 monoclonal antibodies are designed to prevent the cleavage of C5. A murine monoclonal antibody to human C5, m5G1.1-mAb, was humanized (h5G1.1-mAb) by grafting the antibody's antigen-binding CDR regions onto human antibody-derived framework and constant domains. This antibody is being made available by Alexion Pharmaceuticals, and will be used under their IND.

There will be 15 patients entered (with the goal of 12 evaluable patients) distributed among two treatment groups. Patients will be randomized at a 3 to 1 ratio between h5G1.1-mAb and placebo. Following a screening period of no less than 7 days, a 2 month double-blind, randomized treatment period will commence. Patients will receive an active (h5G1.1-mAb, 8mg/kg) bolus infusion every week X 5, then every 2 weeks X 2, or a placebo bolus infusion every week X 5, then every 2 weeks X 2. All patients will be receiving 7 infusions of h5G1.1-mAb or placebo.

The objective is to determine the safety and tolerability of h5G1.1-mAb and to evaluate the pharmacokinetics and pharmacodynamics of this antibody as well as its efficacy in the target population. Safety will be assessed via the collection of adverse events and the evaluation of pre- and post-treatment laboratory data. Efficacy will be assessed by the change in the manual muscle testing score relative to placebo at 2.25 months (one week following the end of the active treatment period) (primary efficacy value), and the change in the muscle enzyme level, MRI findings, skin examination findings and biopsy, and SF-36 (secondary efficacy values).

ELIGIBILITY:
Patients age greater than or equal to 18 years.

Patients with a diagnosis of definite or probable dermatomyositis by criteria of Bohan et. al., with either active rash typical of dermatomyositis, history of rash typical of dermatomyositis, or Gottron's papules.

Patients with a manual muscle testing score less than or equal to 136/170.

Patients with a disease duration greater than or equal to 6 months.

Patients with persistent disease (defined as active rash plus CK greater than or equal to 2 times ULN), or rapidly progressive disease, or response to steroids with inability to taper dose, or unacceptable side effects of steroids.

Patients may be on stable (times 28 days prior to Visit 2) dose of MTX or AZA.

No other immunosuppressive agents times 84 days prior to first dose.

Patients on stable oral steroid use for 28 days prior to Visit 2.

Patients with adequate hematologic function, defined as hemoglobin greater than or equal to 8.5 g/dl, WBC greater than or equal to 3,000 mm(3), neutrophils greater than or equal to 1,200 mm(3), platelets greater than or equal to 100,000 mm(3).

Patients must be willing and able to give informed consent.

Women must be post-menopausal, surgically sterile or practicing a medically approved method of contraception.

Patients with liver disease will be excluded.

Patients with history of alcohol or drug abuse within two years of screening, or a history of positive Hepatitis B or Hepatitis C serology, unless vaccinated will be excluded.

Patients with renal insufficiency, defined as creatinine greater than or equal to 2.0 mg/dl will be excluded.

Patients with history of malignancy, except basal cell carcinoma and remote (greater than or equal to 5 years) malignancies in complete remission will be excluded.

Patients with history of poorly controlled diabetes will be excluded.

Patients with presence or suspicion of active infection, recent serious infection, or chronic/recurrent viral or bacterial infection will be excluded.

Patients with throat culture positive for pathogenic Neisseria species (meningitidis or gonorrhoeae) will be exluded. Subjects with a positive culture may be treated with appropriate antibiotic therapy and retested.

Patients with joint disease or replacement that would interfere with patient's ability to perform muscle testing will be excluded.

Patients with any clinically significant medical condition that is likely to interfere with the participation in the study or the evaluation of the study medication's safety profile will be excluded.

No patients with known or suspected hereditary complement deficiency will be excluded.

Patients with history of allergic reaction to murine proteins will be excluded.

Patients participating in any other investigational drug trial, or exposure to other investigational agent or device within thirty days prior to screening will be excluded.

Pregnant or breastfeeding patients will be excluded.

Women intending to conceive during the course of the study, including follow-up period will be excluded.

Patients with history of HIV, Lyme disease, or other environmentally induced myositis will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17
Dates: Start 2000-04; Study Completion 2001-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Pearson CM, Bohan A. The spectrum of polymyositis and dermatomyositis. Med Clin North Am. 1977 Mar;61(2):439-57. doi: 10.1016/s0025-7125(16)31343-8. No abstract available. PMID 323599
- [Background] Love LA, Leff RL, Fraser DD, Targoff IN, Dalakas M, Plotz PH, Miller FW. A new approach to the classification of idiopathic inflammatory myopathy: myositis-specific autoantibodies define useful homogeneous patient groups. Medicine (Baltimore). 1991 Nov;70(6):360-74. doi: 10.1097/00005792-199111000-00002. PMID 1659647
- [Background] Adams EM, Pucino F, Yarboro C, Hicks JE, Thornton B, McGarvey C, Sonies BC, Bartlett ML, Villalba ML, Fleisher T, Plotz PH. A pilot study: use of fludarabine for refractory dermatomyositis and polymyositis, and examination of endpoint measures. J Rheumatol. 1999 Feb;26(2):352-60. PMID 9972969